CLINICAL TRIAL: NCT03956680
Title: A Phase I Study of BMS-986301 Monotherapy and Combination Therapy With Nivolumab and Ipilimumab in Participants With Advanced Solid Cancers
Brief Title: An Investigational Immunotherapy Study of BMS-986301 Alone or in Combination With Nivolumab, and Ipilimumab in Participants With Advanced Solid Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA046-006; 2018-003610-41 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-05-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Cancers
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A Group 1: BMS-986301 Monotherapy Intramuscular (IM) (Experimental)
  Interventions: Drug: BMS-986301; Biological: Nivolumab; Biological: Ipilimumab
- Part 1A Group 2: BMS-986301 Monotherapy Intratumoral (I-TUMOR) Sub-study (Experimental)
  Interventions: Drug: BMS-986301; Biological: Nivolumab; Biological: Ipilimumab
- Part 1A Group 3: BMS-986301 Monotherapy Intravenous (IV) Sub-study (Experimental)
  Interventions: Drug: BMS-986301; Biological: Nivolumab; Biological: Ipilimumab
- Part 1B Group 4: Systemic BMS-986301 + Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: BMS-986301; Biological: Nivolumab; Biological: Ipilimumab
- Part 1B Group 5: I-TUMOR BMS-986301 + Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: BMS-986301; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Drug: BMS-986301 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: OPDIVO
Biological: Ipilimumab — Specified dose on specified days
  Other Names: YERVOY

SUMMARY:
The main purpose of this study is to characterize the safety, tolerability, dose limiting toxicities, best route of administration, maximum tolerated dose, maximum administered dose, or alternative dose of BMS-986301 alone or in combination with nivolumab and ipilimumab in participants with cancers that have failed to respond to T cell checkpoint inhibiting antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced unresectable/metastatic malignancy of the squamous cell carcinoma of the head and neck (HNSCC), non-small cell lung cancer (NSCLC), melanoma, renal cell carcinoma (RCC), triple negative breast cancer (TNBC), and urothelial carcinoma (UCC), that are refractory to or intolerant of existing therapy(ies) known to provide clinical benefit for the condition of the participant
* Must have experienced radiographically documented progressive disease on or after the most recent therapy
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Women and men must agree to follow specific methods of contraception, if applicable, while participating in the trial

Exclusion Criteria:

* Primary central nervous system (CNS) malignancy
* Other active malignancy requiring concurrent intervention
* Uncontrolled or significant cardiovascular disease

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLTs) | Cycle 1 (28 days)
Incidence of adverse events (AEs) | From Baseline until study exit (up to approximately 2 years)
Incidence of serious adverse events (SAEs) | From Baseline until study exit (up to approximately 2 years)
Incidence of AEs leading to discontinuation | From Baseline until study exit (up to approximately 2 years)
Incidence of deaths | From Baseline until study exit (up to approximately 2 years)
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | From Baseline until disease progression (approximately 2 years)
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | From Baseline until disease progression (approximately 2 years)
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | From Baseline until disease progression (approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (4):
  - Local Institution - 0003, Chicago, Illinois
  - Local Institution - 0005, St Louis, Missouri
  - Local Institution - 0006, Pittsburgh, Pennsylvania
  - Local Institution - 0002, Nashville, Tennessee
- Local Institution - 0001, Toronto, Ontario, Canada

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com